CLINICAL TRIAL: NCT03859362
Title: Pharmacodynamics of Ertapenem in Patients With Urosepsis
Brief Title: Ertapenem in Patients With Urosepsis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Sutep Jaruratanasirikul, Principle Investigator, Prince of Songkla University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ERTAESBL58372141
Record Dates: First submitted 2019-02-25; First posted 2019-03-01 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Patients With Urosepis and Received Ertapenem for Treatment
Keywords: pharmacokinetic, pharmacodynamic, ertapenem, urosepsis
MeSH Terms: interventions — Ertapenem

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ertapenem in urosepsis (Experimental): Ertapenem PK studies were carried out on the 3rd dose of ertapenem administration. Blood samples (3 mL) were obtained by direct venipuncture at the following times: shortly before (time zero) and 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12 and 24 h after the start of ertapenem administration. All blood samples were added to a heparinized tube and centrifuged at 1,000 g for 10 min at 4°C within 5 min.
  Interventions: Drug: Ertapenem Injection

INTERVENTIONS:
Drug: Ertapenem Injection — 1 g of ertapenem q24h, 30 min infusion

SUMMARY:
Ertapenem, a broad-spectrum carbapenem antibiotic, has shown promising in vitro activity agenst ESBL-producing Enterobacteriacae. This agent was licensed in United State of America and Europe for several clinical use in complicated intraabdominal infections, complicated skin and skin-structure infections, acute pelvic infections, complicated urinary tract infections and community-acquired pneumonia. In common with other beta-lactams, ertapenem exhibits primarily time-dependent activity, and the percentage of the exposure time during which the free drug concentration remain above the MIC (%T>MIC) is the pharmacokinetic/pharmacodynamics (PK/PD) index that best correlates with efficacy. Pathophysiological changes in critically ill patients with severe infections resulting in altered PK patterns that may affect therapeutic plasma concentrations and achievement of PD have been found with several antimicrobial agents. The aim of the study was to determine the PK of ertapenem in patients with urosepsis.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age
* Diagnosis of urosepsis

Exclusion Criteria:

* They were pregnant
* Circulatory shock (defined as a systolic blood pressure of < 90 mmHg and pour tissue perfusion)
* Documented hypersensitivity to carbapenems
* Estimated creatinine clearance (CLcr) (determined by the Crockcroft-Goult method) of < 30 mL/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-01 (Actual); Primary Completion 2018-12-30 (Actual); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Concentration of ertapenem in plasma | 48 hours after the ertapenem dose

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Department of Medicine, Faculty of Medicine, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand